CLINICAL TRIAL: NCT04103905
Title: A Multi-Center, Open Label, Single Arm, Multiple Dose Study to Assess the Tolerability，Pharmacokinetics and Efficacy of MIL62 in Chinese Patients With Relapsed/Refractory CD20+ Malignant B-cell Lymphomas
Brief Title: A Study of MIL62 in Treatment of CD20 Positive B-cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIL62-CT01
Record Dates: First submitted 2019-09-18; First posted 2019-09-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2019-08

CONDITIONS: CD20-positive B Cell Non-Hodgkin Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MIL62 (Experimental)
  Interventions: Drug: Recombinant Humanized Monoclonal Antibody MIL62 Injection

INTERVENTIONS:
Drug: Recombinant Humanized Monoclonal Antibody MIL62 Injection — The patients confirming to the eligibility criteria will be assigned to the 5 dose groups (200mg, 400mg, 800mg, 1000mg, and 1500mg, respectively) based on the sequence of inclusion. Each patient received an intravenous infusion of MIL62 on Days 1, 8, and 15 of Cycle 1 and on Day 1 of Cycles 2-8 for a maximum of 8 cycles and 10 infusions. Each cycle was 21 days.

SUMMARY:
This open-label, multicenter,dose-escalating phase I study was designed to evaluate the safety, tolerability, pharmacokinetics and efficacy of MIL62 in Chinese patients with relapsed/refractory CD20-positive B-cell non-Hodgkin lymphoma(NHL) for whom no treatment of higher priority was available.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, >=18 years of age;
2. Diagnosis of Refractory/relapsed CD20+ B-cell lymphoma or B-CLL
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Life expectancy >6 months
5. Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 2 months after discontinuation of all study treatments
6. Able and willing to provide written informed consent and to comply with the study protocol

Exclusion Criteria:

1. Prior use of any investigational antibody therapy within 3 months of study start
2. Prior use of any anti-cancer vaccine
3. Prior administration of radioimmunotherapy 3 months prior to study entry
4. Central nervous system lymphoma
5. History of other malignancy
6. Evidence of significant, uncontrolled concomitant disease
7. Abnormal laboratory values
8. Patients with progressive multifocalleukoencephalopathy (PML)
9. Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C(including HBsAg,HBcAb positive with abnormal HBV DAN or HCV RNA )
10. Known severe allergic reaction or/and infusion reaction to monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced a Dose-limiting Toxicity in Dose Escalation Period of the Study | Baseline to 28 days after the first infusion of MIL62 of the last participant in dose escalation period

SECONDARY OUTCOMES:
Percentage of Participants With Best Overall Response | by the end of Cycle 8 (each cycle is 28 days)
Maximum Observed Plasma Concentration (Cmax) Under Steady State of MIL62 | by the end of Cycle 4 (each cycle is 28 days)
Area Under the Plasma Concentration Versus Time Curve (AUC) of MIL62 Under Steady State | by the end of Cycle 4 (each cycle is 28 days)
Systemic Clearance of MIL62 Under Steady State | by the end of Cycle 4 (each cycle is 28 days)
Volume of Distribution Under Steady State (Vss) of MIL62 | by the end of Cycle 4 (each cycle is 28 days)
Terminal Plasma Half-Life (t1/2) of MIL62 Under Steady State | by the end of Cycle 4 (each cycle is 28 days)
Change in Cluster of Differentiation 19 (CD19+) B Cells | by the end of Cycle 4 (each cycle is 28 days)
Change in Cluster of Differentiation 20 (CD20+) B Cells | by the end of Cycle 4 (each cycle is 28 days)
Percentage of Participants with Positive Anti-Drug Antibodies to MIL62 | by the end of Cycle 4 (each cycle is 28 days)
Progression-free Survival (PFS) in the Study | by the end of the follow-up period of the study
Overall Survival (OS) in the Study | by the end of the follow-up period of the study
Duration of response (DoR) | by the end of the follow-up period of the study
Disease control rate (DCR) | by the end of the follow-up period of the study
Participants With Event-Free Survival (EFS) | by the end of the follow-up period of the study

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Chinese Academy of Medical Sciences (CAMS) & Peking Union Medical College (PUMC)
Locations (1):
- Chinese Academy of Medical Sciences (CAMS) & Peking Union Medical College (PUMC), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No